CLINICAL TRIAL: NCT05914233
Title: Revolutionary Non-Invasive Ultrasound Technology for Vision Restoration in Age-Related Macular Degeneration (AMD) and Retinitis Pigmentosa (RP) Patients
Brief Title: Non-invasive Ultrasound Retinal Stimulation for Vision Restoration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Qifa Zhou, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-23-00143
Record Dates: First submitted 2023-05-08; First posted 2023-06-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration; Retinitis Pigmentosa; Ultrasound Therapy; Complications
Keywords: Ultrasound Stimulation; Retinal; Retinitis pigmentosa; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Tremendous development has been achieved in the matrix ultrasound transducer. The investigators build the signal element ultrasound transducer to provide a stable energy release to stimulate a particular area. The investigators can limit the ultrasound focus to a minor point. The neuron activities induced by the focused 3 Megahertz (MHz) transducers have shown a spatial resolution of 250±50 µm. According to previous study, the Intensity Spatial-Peak Pulse-Average (ISPPA.3) is 26 (Under FDA suggestion of 28).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Stimulation of the ultrasound retinal stimulation Device
  Interventions: Device: Non-invasive ultrasound retinal stimulation Device

INTERVENTIONS:
Device: Non-invasive ultrasound retinal stimulation Device — Record user feelings during the device is working

SUMMARY:
This clinical trial aims to test the safety and feasibility of using a non-invasive ultrasound device to stimulate retinal nerve cells and restore vision in patients with age-related macular degeneration. Previous studies have shown that artificial stimulation, such as electric and optic stimulations, can partially restore vision, but these methods are invasive and pose surgical risks. The study aims to develop a non-invasive method for retinal stimulation. The investigators will follow the FDA guidelines to limit the ultrasound power and adhere to all clinical trial regulations to ensure all participants' safety.

The main questions the investigators aim to answer are:

* Is using high-frequency ultrasound safe using a wearable device for localized retinal neural activity stimulation?
* Does the stimulation through the device restore vision in patients with age-related macular degeneration?

Participants in this study will be asked to undergo Optical Coherence Tomography (OCT) scanning before and after the ultrasound stimulation to evaluate the device's safety. Then, they will receive five stimulation-rest cycles and complete a questionnaire to report what they see and how they feel during the device's operation.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the efficacy and safety of a new non-invasive ultrasound retinal stimulation device for vision restoration in patients with age-related macular degeneration. The investigators will take the following measures:

* The study population will consist of patients with age-related macular degeneration for whom traditional medical treatments have been ineffective and for whom there are no other viable treatment options.
* The investigators will follow the FDA guidelines and adhere to all regulations related to clinical trials to ensure the safety of all participants.
* The investigators will obtain informed consent from each participant and ensure that they fully understand the risks and benefits of the study before enrolling.
* The investigators will closely monitor each participant during the study and record any adverse events or complications.
* The investigators will use high-frequency ultrasound for localized stimulation, which is safe and effective in other studies.

Participants will receive stimulation from the non-invasive ultrasound device for five cycles and complete a questionnaire about their experiences. The researchers will analyze the results to determine the efficacy and safety of the device.

With these measures in place, The investigators believe that the study design and methodology are appropriate and will result in a low-risk study that meets the FDA's requirements for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AMD (regardless of stage and type) or RP. At least two volunteers should diagnose with RP.
2. Age 18 years or older
3. No other eye-related health conditions
4. No allergic history to commercial ultrasound gel
5. Must be willing and able to comply with the protocol testing

Exclusion Criteria:

1. Declining to participate and inability to give informed consent.
2. Unable to comply with the process of the research
3. If the volunteer has optic nerve disease, including the history of glaucoma, optic neuropathy, or other confirmed damage to optic nerve or visual cortex damage
4. Unable to fixate that hinders obtaining high-quality imaging
5. High myopia; refractive error of six diopters and above
6. Pregnancy
7. Subject is participating in another investigational drug or device study that may conflict with the objectives, follow-up, or testing of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2027-01-10 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual function-Assessed by Questionnaire | 2 hours (average duration of procedure)
  A questionnaire will be given to participants. The answers will be recorded as "No" or "Yes." If "Yes" is selected as the participant's answer, their descriptions according to the given questions will be recorded in detail.
Adverse Event | From time of procedure up to 2 hours after process completion
  The nature and number of Treatment-Related Adverse Events.

SECONDARY OUTCOMES:
Comfort Level-Assessed by Questionnaire | 2 hours (average duration of procedure)
  A scale of 0 to 5 will be provided to the participants. 0 is no feeling, and 5 is very pain or uncomfortable

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Zhou, PhD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye J, Tang S, Meng L, Li X, Wen X, Chen S, Niu L, Li X, Qiu W, Hu H, Jiang M, Shang S, Shu Q, Zheng H, Duan S, Li Y. Ultrasonic Control of Neural Activity through Activation of the Mechanosensitive Channel MscL. Nano Lett. 2018 Jul 11;18(7):4148-4155. doi: 10.1021/acs.nanolett.8b00935. Epub 2018 Jun 19. PMID 29916253
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Chaumet-Riffaud AE, Chaumet-Riffaud P, Cariou A, Devisme C, Audo I, Sahel JA, Mohand-Said S. Impact of Retinitis Pigmentosa on Quality of Life, Mental Health, and Employment Among Young Adults. Am J Ophthalmol. 2017 May;177:169-174. doi: 10.1016/j.ajo.2017.02.016. Epub 2017 Feb 22. PMID 28237413
- [Background] Brandolin P, Martinelli G, Zanoni A. [Possibilities of use of neuroleptoanalgesic drugs of type II (dehydrobenzoperidol and fentanyl) in emergency abdominal surgery in aged patients]. Acta Anaesthesiol. 1968;19:Suppl 4:93+. No abstract available. Italian. PMID 5757022
- [Background] Chou R, Dana T, Bougatsos C, Grusing S, Blazina I. Screening for Impaired Visual Acuity in Older Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2016 Mar 1;315(9):915-33. doi: 10.1001/jama.2016.0783. PMID 26934261
- [Background] TASSICKER GE. Preliminary report on a retinal stimulator. Br J Physiol Opt. 1956 Apr;13(2):102-5. No abstract available. PMID 13315967
- [Background] Humayun MS, Weiland JD, Fujii GY, Greenberg R, Williamson R, Little J, Mech B, Cimmarusti V, Van Boemel G, Dagnelie G, de Juan E. Visual perception in a blind subject with a chronic microelectronic retinal prosthesis. Vision Res. 2003 Nov;43(24):2573-81. doi: 10.1016/s0042-6989(03)00457-7. PMID 13129543
- [Background] Ahuja AK, Dorn JD, Caspi A, McMahon MJ, Dagnelie G, Dacruz L, Stanga P, Humayun MS, Greenberg RJ; Argus II Study Group. Blind subjects implanted with the Argus II retinal prosthesis are able to improve performance in a spatial-motor task. Br J Ophthalmol. 2011 Apr;95(4):539-43. doi: 10.1136/bjo.2010.179622. Epub 2010 Sep 29. PMID 20881025
- [Background] da Cruz L, Dorn JD, Humayun MS, Dagnelie G, Handa J, Barale PO, Sahel JA, Stanga PE, Hafezi F, Safran AB, Salzmann J, Santos A, Birch D, Spencer R, Cideciyan AV, de Juan E, Duncan JL, Eliott D, Fawzi A, Olmos de Koo LC, Ho AC, Brown G, Haller J, Regillo C, Del Priore LV, Arditi A, Greenberg RJ; Argus II Study Group. Five-Year Safety and Performance Results from the Argus II Retinal Prosthesis System Clinical Trial. Ophthalmology. 2016 Oct;123(10):2248-54. doi: 10.1016/j.ophtha.2016.06.049. Epub 2016 Jul 21. PMID 27453256
- [Background] Lu Y, Brommer B, Tian X, Krishnan A, Meer M, Wang C, Vera DL, Zeng Q, Yu D, Bonkowski MS, Yang JH, Zhou S, Hoffmann EM, Karg MM, Schultz MB, Kane AE, Davidsohn N, Korobkina E, Chwalek K, Rajman LA, Church GM, Hochedlinger K, Gladyshev VN, Horvath S, Levine ME, Gregory-Ksander MS, Ksander BR, He Z, Sinclair DA. Reprogramming to recover youthful epigenetic information and restore vision. Nature. 2020 Dec;588(7836):124-129. doi: 10.1038/s41586-020-2975-4. Epub 2020 Dec 2. PMID 33268865
- [Background] Fomenko A, Neudorfer C, Dallapiazza RF, Kalia SK, Lozano AM. Low-intensity ultrasound neuromodulation: An overview of mechanisms and emerging human applications. Brain Stimul. 2018 Nov-Dec;11(6):1209-1217. doi: 10.1016/j.brs.2018.08.013. Epub 2018 Aug 23. PMID 30166265
- [Background] Liu SH, Lai YL, Chen BL, Yang FY. Ultrasound Enhances the Expression of Brain-Derived Neurotrophic Factor in Astrocyte Through Activation of TrkB-Akt and Calcium-CaMK Signaling Pathways. Cereb Cortex. 2017 Jun 1;27(6):3152-3160. doi: 10.1093/cercor/bhw169. PMID 27252349
- [Background] Chen Y, Shi Z, Shen Y. Eye damage due to cosmetic ultrasound treatment: a case report. BMC Ophthalmol. 2018 Aug 29;18(1):214. doi: 10.1186/s12886-018-0891-2. PMID 30157786
- [Result] Lu G, Qian X, Gong C, Ji J, Thomas BB, Humayun MS, Zhou Q. Ultrasound Retinal Stimulation: A Mini-Review of Recent Developments. IEEE Trans Ultrason Ferroelectr Freq Control. 2022 Dec;69(12):3224-3231. doi: 10.1109/TUFFC.2022.3220568. Epub 2022 Nov 24. PMID 36343006
- See also: Noninvasive Ultrasound Retinal Stimulation for Vision Restoration at High Spatiotemporal Resolution — https://pubmed.ncbi.nlm.nih.gov/37850175/